CLINICAL TRIAL: NCT02728726
Title: Randomized Double---Blinded, Controlled Trial to Compare the Effectiveness of Sugammadex vs. Placebo to Prevent Residual Neuromuscular Block in the Post---Anesthesia Care Unit as Evaluated With a Non---Invasive Respiratory Volume Monitor
Brief Title: Sugammadex vs Placebo to Prevent Residual Neuromuscular Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); University of Texas (Other); Respiratory Motion, Inc. (Industry)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-008685; NCT02822001 (obsolete NCT alias)
Record Dates: First submitted 2016-03-15; First posted 2016-04-05 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: General Surgery
Keywords: Postoperative respiratory depression; Neuromuscular Agents
MeSH Terms: interventions — Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sugammadex (Experimental): Subjects will have Sugammadex administered after routine reversal of anesthesia is performed and patient is extubated.
  Interventions: Drug: Sugammadex
- Placebo (Placebo Comparator): Subjects will have Placebo administered after routine reversal of anesthesia is performed and patient is extubated.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sugammadex — Sugammadex will be administered intravenously at 2 mg/kg after routine reversal of anesthesia is performed and subject is extubated.
  Other Names: Bridion
  Arms: Sugammadex
Drug: Placebo — Placebo will be administered intravenously at 2 mg/kg after routine reversal of anesthesia is performed and subject is extubated.
  Arms: Placebo

SUMMARY:
The study is designed to determine whether patients who receive sugammadex immediately after tracheal extubation will exhibit a decrease in the incidence of postoperative residual paralysis and an associated decrease in the incidence of postoperative respiratory depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery with general anesthesia
* Patients weighing > or = 80 pounds
* Patients not intubated prior to surgery
* Patients who are able to give informed consent

Exclusion Criteria:

* Patients unable to give informed consent.
* Patients whose condition will not allow for placement of the electrode PadSet of ExSpiron
* Patients who are anticipated to remain intubated in recovery period.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Florida, Jacksonville, Florida
  - The University of Texas, UTHealth, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugammadex: Subjects had Sugammadex administered after routine reversal of anesthesia was performed and subject was extubated.
  Sugammadex: Sugammadex administered intravenously at 2 mg/kg after routine reversal of anesthesia was performed and subject was extubated.
- Placebo: Subjects had Placebo administered after routine reversal of anesthesia was performed and subject was extubated.
  Placebo: Placebo was administered intravenously at 2 mg/kg after routine reversal of anesthesia was performed and subject was extubated.
Period: Overall Study
Arm/Group | Sugammadex | Placebo
Started | 127 | 133
Completed | 127 | 133
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugammadex | Placebo | Total
Number analyzed (Participants) | 127 | 133 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.65 (16.74) | 52.13 (16.07) | 52.87 (16.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 37 | 82
  Male | 82 | 96 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Baseline race/ethnicity was not collect or provided for 57 subjects in the Sugammadex arm. Baseline race/ethnicity was not collect or provided for 59 subjects in the Placebo arm. Could not use Race (NIH/OMB) pre-structured Baseline Measure, as there is not a Hispanic or Latino in that option.
  Participants
    American Indian or Alaska Native: number analyzed (Participants) | 70 | 74 | 144
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 2 | 2
    Native Hawiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 5 | 4 | 9
    White | 61 | 67 | 128
    Hispanic or Latino | 1 | 1 | 2
    More than one race | 0 | 0 | 0
    Unknown | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 127 | 133 | 260

OUTCOME MEASURES:

1. Primary Outcome: Decreased Minute Ventilation (MV)
Description: The number of subjects who have a MV as defined as [MV <80% MV predicted (MVPRED) based on Body Surface Area]. MV (or respiratory minute volume or minute volume) is the volume of gas inhaled (inhaled minute volume) or exhaled (exhaled minute volume) from a person's lungs per minute.
Time Frame: 15---30 minutes after Post-anesthesia care unit (PACU) arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 62 | 54
Participants | 20 | 26

2. Primary Outcome: Decreased Average Minute Ventilation (MV)
Description: The number of subjects who have an average MV <80% MV predicted (MVPRED) based on Body Surface Area. MV (or respiratory minute volume or minute volume) is the volume of gas inhaled (inhaled minute volume) or exhaled (exhaled minute volume) from a person's lungs per minute.
Time Frame: 15---30 minutes after Post-anesthesia care unit (PACU) arrival
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 62 | 54
Participants | 20 | 26

3. Secondary Outcome: Train of Four (TOF) Ratio
Description: The number of subjects to have a normal TOF ratio (>0.90) indicative of full neuromuscular recovery in the Post-anesthesia care unit (PACU)
Time Frame: upon PACU discharge, approximately 8 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Sugammadex | Placebo
Number analyzed (Participants) | 62 | 54
Participants | 42 | 29

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from baseline to end of study (discharged from the recovery room), approximately 8 hours
Arm/Group | Sugammadex | Placebo
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/133
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/133
Other Adverse Events (participants affected / at risk) | 0/127 | 2/133
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sugammadex (N=127) | Placebo (N=133)
Cardiac Catherization post surgery - Stent placed (Cardiac disorders) | 0 | 1
Extended intubation (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/26/NCT02728726/Prot_SAP_000.pdf